CLINICAL TRIAL: NCT02154711
Title: Magnetic Resonance Imaging (MRI) Muscle Phenotyping in Mitochondrial Disease
Status: Completed | Type: Observational
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Shana McCormack, Instructor in Pediatrics, University of Pennsylvania
Other Study IDs: 819440
Record Dates: First submitted 2014-05-29; First posted 2014-06-03 (Estimated); Last update posted 2024-08-29 (Actual); Status verified 2024-08

CONDITIONS: Mitochondrial Disease
Keywords: mitochondrial disease; magnetic resonance imaging; magnetic resonance spectroscopy; creatine; phosphocreatine
MeSH Terms: conditions — Mitochondrial Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Mitochondrial Disease: Individuals with genetic diagnoses (nuclear or mitochondrial) of mitochondrial disease
- Unaffected: Healthy individuals, without mitochondrial disease

SUMMARY:
The purpose of the study is to use a new research imaging technique, a kind of magnetic resonance imaging (MRI), to measure important metabolic features of muscle, including mitochondrial function, in people with mitochondrial disease and in healthy individuals. (Mitochondria are tiny organelles that generate energy for the body.)

It is hoped that this new strategy will help physicians to understand better the health problems of people with mitochondrial disease. Eventually, this could lead to better diagnostic and treatment approaches.

DETAILED DESCRIPTION:
There are two study-related visits.

The first visit is a "screening" visit to ensure eligibility. This includes fasting blood tests. The second visit is an MRI scanning session. This also takes around 2 - 3 hours, with no more than 1.5 hours spent in the actual MRI machine. It may be possible to complete these two visits on the same day. Otherwise, the MRI session should occur within 3 months of the screening visit. In addition, an optional physical capacity visit will occur on the same day as the MRI session.

ELIGIBILITY:
Group 1) Mitochondrial Disease:

Inclusion Criteria:

* Genetic diagnosis of mitochondrial disease
* Be able to perform sub-maximal leg exercise for several minutes
* Be able to provide written, informed consent
* Cognitively and medically stable and able to comply with study procedures
* Able to fast for 4 hours prior to blood draw and/or MRI scanning
* Be willing to stop taking any over-the-counter vitamins and supplements that are neither prescribed nor recommend by their physician for 2 weeks prior to MRI scanning

Exclusion Criteria:

* Diabetes
* Alcohol/substance abuse
* Smoking
* Use of any investigational agents within 4 weeks of enrollment
* Any contraindication to MRI scanning

Group 2) Healthy Individuals:

Inclusion Criteria:

* Be able to perform sub-maximal leg exercise for several minutes
* Be able to provide written, informed consent
* Cognitively and medically stable and able to comply with study procedures
* Able to fast for 4 hours prior to blood draw and/or MRI scanning
* Be willing to stop taking any over-the-counter vitamins and supplements that are neither prescribed nor recommend by their physician for 2 weeks prior to MRI scanning

Exclusion Criteria:

* Carry a diagnosis of mitochondrial disease
* Have a first-degree relative with a diagnosis of mitochondrial disease
* Diabetes
* Alcohol/substance abuse
* Smoking
* Use of any investigational agents within 4 weeks of enrollment
* Any contraindication to MRI scanning

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Two groups of subjects: 1) mitochondrial disease and 2) healthy individuals
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2014-05; Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Creatine Recovery Time | 15 minutes

SECONDARY OUTCOMES:
Phosphocreatine recovery time | 15 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Shana E McCormack, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States